CLINICAL TRIAL: NCT06817486
Title: The Effects of Mornıng and Evenıng Runnıng on Respıratory Functıon and Lower Extremıty Strength in Pre-Adolescent Male Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coşkun YILMAZ (Other)
Responsible Party: Sponsor-Investigator, Coşkun YILMAZ, Sports Scientist ASSOC. PROF., Gümüşhane Universıty
Organization: Gümüşhane Universıty (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: E-95674917-108.99-239802; E-95674917-108.99-239802 (Other: GUMUSHANE UNIVERSITY)
Record Dates: First submitted 2025-01-27; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: HEALTHY PREADOLESCENT MALE; Effects of Running on Daily Variation in Healthy Adolescent Children
Keywords: Lower extremity, respiratory function, children, physical activity, lifestyle; Healthy preadolescent children
MeSH Terms: conditions — Respiratory Aspiration; Motor Activity

STUDY DESIGN:
Intervention Model Description: In our study, participants were grouped into 'moderate and definite morning type' (MRG, n=25), 'no type' (CON, n=25) and 'moderate and definite evening type' (ERG, n=25) according to their responses to the questionnaire assessing morning/evening status.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MORNİNG RUNNİNG (Experimental): TRAİNİNG
  Interventions: Other: RUNNİNG TRAİNİNG; Procedure: TRAİNİNG
- EVENİNG RUNİNG (Experimental): TRAİNİNG
  Interventions: Other: RUNNİNG TRAİNİNG; Procedure: TRAİNİNG
- CONTROL (No Intervention): No ıntervention

INTERVENTIONS:
Other: RUNNİNG TRAİNİNG — Running training It was performed between 08:00 and 10:00 for morning running and between 18:00 and 20:00 for evening running (Bessot et al., 2014). The exercise intensity of each child in the running group was determined as the 50% heart rate (HR) according to the Karvonen formula (target pulse: (220-age-basal pulse) × intensity) + basal pulse). HR was determined via a telemetric heart rate monitor (PolarM400, Finland) during the first week of running training. Environmental conditions are known to influence the degree of airway epithelial disruption during high-intensity exercise (Boukelia et al., 2017). Therefore, all the participants performed continuous running exercise on a football field in Kelkit/Gümüşhane/Turkey (altitude: 1373 m). It was performed for 50 minutes (including 10 min warm-up and cool-down), 3 days a week, for 8 weeks at the set target heart rate. Each session was supervised by trainers. Running included approximately 10 minutes of warm-up and cool-down with stati
  Arms: EVENİNG RUNİNG; MORNİNG RUNNİNG
Procedure: TRAİNİNG — RUNNING TRAINING WAS DONE
  Arms: EVENİNG RUNİNG; MORNİNG RUNNİNG

SUMMARY:
The objective of this study was to examine the impact of eight weeks of morning and evening running on lower extremity strength and respiratory function in 10-12-year-old male soccer players. The participants visited the laboratory 3 times with 1-day intervals before and after the training. The measurements included maximal inspiratory pressure (MIP), maximal expiratory pressure (MEP), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and the FEV1/FVC ratio, agility and functional performance tests (FPTs) for the dominant and nondominant legs. The results of investigators study indicated that morning running was more effective than other forms of exercise in developing the respiratory system. The greatest improvement in FVC, FEV1, MIP, and MEP values was observed in those who performed morning runs (p< 0.001). The findings of our study indicate that morning running is more effective than running the dominant leg in a series of lower extremity strength tests, including the single leg (SL) and triple leg (THD) crossover hop for distance tests (CHDs) and the 6 m timed-hop test (6 m THT). The results were statistically significant (p=0.000). With respect to the nondominant leg, the SL and 6-meter THT tests were more effective in the morning running group than in the evening running group (p=0.000). The morning running group had better agility performance than the evening and control groups did. As a result, it was determined that morning jogging had a positive effect on respiratory muscle strength, respiratory function and lower extremity strength in children.

DETAILED DESCRIPTION:
The Effects of Mornıng and Evenıng Runnıng on Respıratory Functıon and Lower Extremıty Strength in Pre-Adolescent Male Footballers Coşkun YILMAZ, Süreyya Yonca SEZER, Özgür EKEN, Baha Engin Çelikel ABSTRACT The objective of this study was to examine the impact of eight weeks of morning and evening running on lower extremity strength and respiratory function in 10-12-year-old male soccer players. The participants visited the laboratory 3 times with 1-day intervals before and after the training. The measurements included maximal inspiratory pressure (MIP), maximal expiratory pressure (MEP), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and the FEV1/FVC ratio, agility and functional performance tests (FPTs) for the dominant and nondominant legs. The results of our study indicated that morning running was more effective than other forms of exercise in developing the respiratory system. The greatest improvement in FVC, FEV1, MIP, and MEP values was observed in those who performed morning runs (p< 0.001). The findings of investigators study indicate that morning running is more effective than running the dominant leg in a series of lower extremity strength tests, including the single leg (SL) and triple leg (THD) crossover hop for distance tests (CHDs) and the 6 m timed-hop test (6 m THT). The results were statistically significant (p=0.000). With respect to the nondominant leg, the SL and 6-meter THT tests were more effective in the morning running group than in the evening running group (p=0.000). The morning running group had better agility performance than the evening and control groups did. As a result, it was determined that morning jogging had a positive effect on respiratory muscle strength, respiratory function and lower extremity strength in children.

Keywords: Lower extremity, respiratory function, children, physical activity, lifestyle Introduction Several studies have focused on elucidating the impact of homeostatic alterations on athletic performance across the diurnal cycle. These investigations have consistently demonstrated that athletes exhibit considerable discrepancies in their performance, contingent on the temporal occurrence of their exercise regimen. In these processes, known as circadian rhythm, previous studies have reported a positive effect of evening training on sporting performance compared with training in the morning.

It has been demonstrated that long-term combined strength and endurance training in the evening can result in greater increases in muscle hypertrophy and mass than training conducted in the morning. These findings have been consistently observed in cardiovascular fitness tests, such as swimming and cycling, and in strength tests, such as standing vertical jumps (countermovement jumps) and isometric muscle contractions. This variation in athletic performance is strongly associated with the mechanisms of circadian rhythm. Consequently, the circadian rhythm represents a crucial consideration in the development of training regimens.

The study of circadian rhythms, defined as the cyclic 24-hour patterns of physiological functions, including lung function, has emerged as a prominent area of interest in both basic and clinical research. The maintenance of circadian rhythms is regulated by the 'circadian clock', which is located in the suprachiasmatic nucleus of the hypothalamus. This process is organized by the hypothalamic-pituitary axis, the autonomic nervous system and clock proteins that form regulatory feedback loops. The suprachiasmatic nucleus in the hypothalamus serves as the primary circadian clock, generating these rhythms. It is synchronized with external cues, including light-dark cycles, mealtimes and social interactions. Furthermore, it regulates rhythmic changes in human physiology and coordinates the timing of processes such as the sleep-wake cycle, fluctuating activity levels and the synchronization of skeletal muscle functionality. Numerous factors related to circadian rhythm (body temperature, chronotype (morning type vs. evening type), training programs and daily fluctuations in biochemical markers) have been shown to contribute to diurnal variation in athletic performance. The presence of a circadian rhythm in lung function, which is one of these factors, is also known.

The capacity of the lungs to regulate oxygen intake during running is a key factor in both running economy and performance. It has been demonstrated in the literature that regular running training has a significant effect on performance peaks, with the greatest benefits observed when training is conducted in the morning. Additionally, when training is performed in the afternoon or evening, it has been shown to increase the amplitude of daily variations at the neuromuscular level. In the context of professional marathon running, evidence suggests that prioritizing morning training sessions may lead to enhanced performance outcomes. In the literature, running training, in which circadian rhythm is taken into account, is generally performed on adult and young athletes, but there are no studies on how morning running and evening running affect lower extremity strength and respiratory functions in studies on child athletes. Therefore, this study aimed to determine the effects of 8 weeks of morning running and evening running on lower extremity strength and respiratory function in 10-12-year-old male football players. It is hypothesized that the data obtained from morning and evening running training differ. This information may prove useful to coaches and sports scientists engaged in the design of training programmes in their professional capacities.

Materials and methods Research Design and Sampling Procedure In this study, a parallel two-group pre-test-post-test randomized controlled trial was conducted according to CONSORT guidelines. All participants and their parents were given detailed information about before the study, and written informed consent was obtained in accordance with the ethical principles described in the Declaration of Helsinki. Help was received from a 3rd-level athleticism coach for planning and implementing running exercises to be used in the project. The study was designed according to the rules of the Declaration of Helsinki and approved by the ethics committee for scientific research of Gümüşhane University (at its meeting on 21.02.24 and number 2024/2; decision number E-95674917-108.99-239802).

Experimental design The participants were visited the laboratory on three occasions, at one-day intervals prior to and following the training period. During the initial visit, the participants and their parents were furnished with comprehensive information regarding the test and pilot tests were administered to the participants.In the second visit, respiratory function tests were conducted, and measurements of respiratory muscle strength, height and body weight were taken.In the third and final visit, the dominant leg was determined, and functional performance tests were performed for the dominant and non-dominant leg. All tests were performed at the same time of day, after the participants were instructed to maintain a normal diet and sleep routine and to avoid intense exercise in the 24 hours prior to testing.Participants fasted for 3 hours before testing and drank 500ml of water 2 hours before testing. All measurements were repeated after eight weeks of running training. During the study, the children were asked to sleep at specific time intervals (9-12 hours) to ensure that their sleep patterns were consistent.

Population and sample The aim of this study was to investigate the effects of morning and evening running training on lower extremity strength, agility performance and respiratory function in 10-12-year-old male soccer players who had been training regularly for at least 2 years. A power analysis was performed via the G.Power 3.1 program to determine the sample size of the study, and the d value was found to be 1.12 (α=0.05, 1-β=0.95, η2p = 0.8). As a result of the analysis, it was decided to include at least 25 participants for each group in the study. The studies were divided into 3 groups: morning running (MRG), evening running (ERG) and a control (CON) groups.

Chronotype The HS-MEQ was used to assess the chronotype of each participant. On the basis of the scores obtained, individuals were classified into one of five chronotype categories: definite evening type (DET) (16--30), moderate evening type (MET) (31--41), no type (NT) (42--58), moderate morning type (MMT) (59--69) and definite morning type (DMT) (70--86). As grouping athletes by chronotype results in significant diurnal variation and better performance data can be obtained when training and testing sessions are circadian in nature, the study grouped athletes by chronotype. In our study, participants were grouped into 'moderate and definite morning type' (MRG, n=25), 'no type' (CON, n=25) and 'moderate and definite evening type' (ERG, n=25) according to their responses to the questionnaire assessing morning/evening status. Participants who answered 'no type' were included in the control group. The reason why extreme chronotypes were not found in the samples in this study was that such chronotypes were not included in the study.

Lower extremity strength tests Dominant and nondominant foot measurements were taken for functional performance tests (FPTs), which were used to determine the subjects' lower extremity strength. Prior to each test, the subjects were instructed on how to perform the measurement. Three trials were performed for each test prior to the actual measurements. After the trial repetitions, the participant was subjected to 3 main tests, and the success criterion in the test was determined as the subject landing on one leg with full stabilization and staying there for three seconds. The subjects rested for 30 seconds between trials. Arm movement was allowed during the movement, and no restrictions were imposed. For all the trials, a 30 cm strip was drawn on the ground as a starting point, a 6 m long and 15 cm wide strip was placed vertically on the ground from the center of this strip, and all the measurements were taken on this platform.

Single Leg Hop for Distance In the TAA test, subjects start standing on one leg at the marked starting line and, when ready, jump horizontally and as far as they can jump so that they fall on the same leg; the result is determined by the successful attempt between the starting line and the subject's heel and recorded in cm.

Triple jump for distance In the UAA test, the subject began by standing on one leg at the start line and, when ready, jumped horizontally as long as he could three times in succession without stopping. The distance between the starting line and the heel height of the subject's fall was recorded in cm.

Single Leg 6 m. Timed Hop Test The subject stands on one foot at the start line and finishes the 6-meter track in the fastest possible time. The test began at the start line and ended when the subject's heel touched the first point at which the subject crossed the finish line. All the subjects were tested three times, with a rest period of 2 minutes between each test. The test was timed in seconds using a standard stopwatch. The best time from the three trials was recorded in seconds. The use of arm movements during movement was allowed, and no restrictions were imposed.

Crossover Hop for Distance The subject stands on one foot at the starting line and performs 3 jumps forward, and the distance jumped is recorded in cm. The first jump starts diagonally opposite the foot used and continues laterally to the side of the fall. For each test, the subjects were given three repetitions. The criterion for success in the test was that the subject landed with full stabilization on the leg and remained standing for three seconds. The best jump distance was recorded in cm. The subjects were given a 30 second rest interval between each trial.

505 Agility test: This test consists of measuring the time taken to complete the last 5 m of a 15 m track. The time within the first 10 m from the start of the test is not included in the test score. When the next 5 m distance is passed for the first time, the recording begins and stops when the same distance is returned.

Measurement of height and weight: A Seca 769 electronic height measuring device (Seca Anonim Şirketi, Hamburg, Germany) was used. The device measures height with an accuracy of 0.1 cm and body weight with an accuracy of 0.01 kg. Body weight was measured in kilograms (kg) without shoes and wearing shorts and a T-shirt to avoid influencing the participants' weight. Height was measured in centimeters (cm) without shoes, with the body weight evenly distributed on both feet.

Pulmonary function tests: FEV1, FEV1/FVC (Tiffenau index), and FVC capacity were analyzed via a CPFS/D USB spirometer from MGF Diagnostics (Saint Paul, Minnesota, USA). Measurements were taken between 15:00 and 17:00 for all participants to obtain the highest spirometric throughput. Participants with FEV1/FVC <75%, any chronic or pulmonary disease, medication that could affect lung function, or a history of upper respiratory tract infection were excluded from the study. Lung function tests were performed with the participants in the standing position. During the tests, the participants wore a nose clip and were instructed to hold their lips tightly around the mouthpiece to prevent air from escaping.

Respiratory muscle strength (measurement of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP)): MIPs and MEPs were measured via a hand-held portable oral pressure meter (MicroRPM, CareFusion Micro Medical, Kent, UK) according to the American Thoracic Society and European Respiratory Society guidelines. With the appropriate filters and holders in place, the nasal airway was closed with a clip. The mouthpiece assembly included a 1 mm hole to prevent glottic closure and minimize the contribution of the buccinator muscles during inspiration. Inspiratory and expiratory maneuvers were performed in the standing position, with MIP and MEP measurements started at the residual volume and total lung capacity, respectively, and continued for at least 1 second. The measurements were repeated until there was a 5% difference between the 2 best results, and the results were recorded as the mean cm H2O.

Running training It was performed between 08:00 and 10:00 for morning running and between 18:00 and 20:00 for evening running. The exercise intensity of each child in the running group was determined as the 50% heart rate (HR) according to the Karvonen formula (target pulse: (220-age-basal pulse) × intensity) + basal pulse). HR was determined via a telemetric heart rate monitor (PolarM400, Finland) during the first week of running training. Environmental conditions are known to influence the degree of airway epithelial disruption during high-intensity Exercise. Therefore, all the participants performed continuous running exercise on a football field in Kelkit/Gümüşhane/Turkey (altitude: 1373 m). It was performed for 50 minutes (including 10 min warm-up and cool-down), 3 days a week, for 8 weeks at the set target heart rate. Each session was supervised by trainers. Running included approximately 10 minutes of warm-up and cool-down with static stretching and light exercises of the relevant muscle groups. The coaches were responsible for monitoring the athletes' running technique and speed, ensuring safety and providing motivation. Both groups were provided sufficient water to avoid dehydration.

Statistical analysis. The research data were analyzed via IBM SPSS Statistics 24. Descriptive data are presented as the means and standard deviations. The normality of the data was examined via the Kolmogorov-Smirnov test, which revealed that the data were normally distributed. For parametric data, the dependent group t test (paired samples t test) was used for within-group, pretest and posttest comparisons, and ANOVA was used for the developmental results obtained with the posttest-pretest = difference formula. Statistical significance was based on a p value of < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Being between 10-12 years old Being healthy Being able to do running training FeV1/FVC <75%

Exclusion Criteria:

* Not being between 10-12 years old Having any disease Not being able to do running training FEV1/FVC >75%

Ages: 10 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
post training | 8 weeks
  After 8 weeks of running training
post training | 8 weeks
  Running training increases respiratory functions, increases respiratory muscle strength, reduces agility score, increases leg strength rates,

CONTACTS AND LOCATIONS:
Locations (1):
- Gumushane Univetsity, Gümüşhane, Kelkit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
THE PERSONAL DATA WILL BE SHARED IF REQUESTED.